CLINICAL TRIAL: NCT00880568
Title: A Phase I Dose Escalation Study of MK1496 in Patients With Advanced Solid Tumor
Brief Title: Phase I Study of MK-1496 in Patients With Advanced Solid Tumor (MK-1496-002 AM 4)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1496-002; 2009_575
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms; Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- MK-1496 20 mg (21-Day Cycle) (Experimental): Participants receiving MK-1496 20 mg on Day 1 of each 21-day cycle
  Interventions: Drug: MK-1496
- MK-1496 40 mg (21-Day Cycle) (Experimental): Participants receiving MK-1496 40 mg on Day 1 of each 21-day cycle
  Interventions: Drug: MK-1496
- MK-1496 80 mg (21-Day Cycle) (Experimental): Participants receiving MK-1496 80 mg on Day 1 of each 21-day cycle
  Interventions: Drug: MK-1496
- MK-1496 120 mg (21-Day Cycle) (Experimental): Participants receiving MK-1496 120 mg on Day 1 of each 21-day cycle
  Interventions: Drug: MK-1496
- MK-1496 20 mg (28-Day Cycle) (Experimental): Participants receiving MK-1496 20 mg on Days 1, 3, 8, 10, 15, and 17 of each 28-day cycle
  Interventions: Drug: MK-1496
- MK-1496 40 mg (28-Day Cycle) (Experimental): Participants receiving MK-1496 40 mg on Days 1, 3, 8, 10, 15, and 17 of each 28-day cycle
  Interventions: Drug: MK-1496
- MK-1496 80 mg (28-Day Cycle) (Experimental): Participants receiving MK-1496 80 mg on Days 1, 3, 8, 10, 15, and 17 of each 28-day cycle
  Interventions: Drug: MK-1496
- MK-1496 100 mg (28-Day Cycle) (Experimental): Participants receiving MK-1496 100 mg on Days 1, 3, 8, 10, 15, and 17 of each 28-day cycle
  Interventions: Drug: MK-1496
- MK-1496 120 mg (28-Day Cycle) (Experimental): Participants receiving MK-1496 120 mg on Days 1, 3, 8, 10, 15, and 17 of each 28-day cycle
  Interventions: Drug: MK-1496

INTERVENTIONS:
Drug: MK-1496 — MK-1496 (20 to 120 mg), orally, administered on Day 1 of each 21-day cycle
  Arms: MK-1496 120 mg (21-Day Cycle); MK-1496 20 mg (21-Day Cycle); MK-1496 40 mg (21-Day Cycle); MK-1496 80 mg (21-Day Cycle)
Drug: MK-1496 — MK-1496 (20 to 120 mg), orally, administered on Days 1 and 3 each week for 3 weeks (Days 1, 3, 8, 10, 15 and 17) of each 28-day cycle
  Arms: MK-1496 100 mg (28-Day Cycle); MK-1496 120 mg (28-Day Cycle); MK-1496 20 mg (28-Day Cycle); MK-1496 40 mg (28-Day Cycle); MK-1496 80 mg (28-Day Cycle)

SUMMARY:
This study determines recommended clinical dose, to evaluate the safety, tolerability and pharmacokinetics of MK-1496 in patients with locally advanced and/or metastatic solid tumors who have failed standard therapy or for whom no standard therapy exists, in two dosing schedules in Japan.

ELIGIBILITY:
Inclusion Criteria

* Participant must have a histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist.
* Participant must have Performance Status 0 or 1.
* Participant must have adequate organ function.

Exclusion Criteria

* Participant has had chemotherapy, radiotherapy, or biological therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to registration.
* Participant has received 4 or greater regimens of chemotherapy (adjuvant therapy and incomplete 1 cycle treatment are not considered as 1 regimen).
* Participant has known hypersensitivity to the components of study drug or its analogs.
* Participant has had prescription or non-prescription drugs or other products known to be moderate or potent inhibitors/inducers of cytochrome P (CYP)3A4, or substrates of CYP3A4 with narrow therapeutic window.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-1496 20 mg (21-Day Cycle) | MK-1496 40 mg (21-Day Cycle) | MK-1496 80 mg (21-Day Cycle) | MK-1496 120 mg (21-Day Cycle) | MK-1496 20 mg (28-Day Cycle) | MK-1496 40 mg (28-Day Cycle) | MK-1496 80 mg (28-Day Cycle) | MK-1496 100 mg (28-Day Cycle) | MK-1496 120 mg (28-Day Cycle)
Started | 3 | 3 | 3 | 1 | 3 | 3 | 6 | 2 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 1 | 3 | 3 | 6 | 2 | 3
Not completed — Disease progression | 3 | 3 | 3 | 1 | 3 | 3 | 5 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1496 20 mg (21-Day Cycle) | MK-1496 40 mg (21-Day Cycle) | MK-1496 80 mg (21-Day Cycle) | MK-1496 120 mg (21-Day Cycle) | MK-1496 20 mg (28-Day Cycle) | MK-1496 40 mg (28-Day Cycle) | MK-1496 80 mg (28-Day Cycle) | MK-1496 100 mg (28-Day Cycle) | MK-1496 120 mg (28-Day Cycle) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 3 | 3 | 6 | 2 | 3 | 27
Age, Continuous [Median (Full Range); unit: Years] | 65.0 [64 to 69] | 57.0 [54 to 71] | 61.0 [53 to 75] | 56.0 [56 to 56] | 52.0 [48 to 63] | 51.0 [43 to 58] | 62.5 [56 to 71] | 57.5 [42 to 73] | 68.0 [59 to 68] | 61.0 [42 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 0 | 2 | 2 | 3 | 2 | 1 | 14
  Male | 2 | 1 | 2 | 1 | 1 | 1 | 3 | 0 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: Dose-limiting toxicities (DLTs) are any adverse events that are not clearly related to disease progression including Grade 4 neutropenia, Grade 3 or 4 febrile neutropenia, thrombocytopenic bleeding or Grade 4 thrombocytopenia, and any Grade 3 or 4 non hematologic toxicity. An adverse event (AE) is any unfavorable and unintended change in the structure and function (Clinical AE) or chemistry (Laboratory AE) of the body temporally associated with the use of study product, whether or not considered related to the use of the product.
Time Frame: Cycle 1 (up to 21 or 28 days, depending on treatment arm)
Population: All participants in the first cycle of each dosing schedule (21 or 28 days)
Measure: Number; unit: participants
Arm/Group | MK-1496 20 mg (21-Day Cycle) | MK-1496 40 mg (21-Day Cycle) | MK-1496 80 mg (21-Day Cycle) | MK-1496 120 mg (21-Day Cycle) | MK-1496 20 mg (28-Day Cycle) | MK-1496 40 mg (28-Day Cycle) | MK-1496 80 mg (28-Day Cycle) | MK-1496 100 mg (28-Day Cycle) | MK-1496 120 mg (28-Day Cycle)
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 3 | 3 | 6 | 2 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

2. Secondary Outcome: Area Under the Curve From Hour 0 to Hour 24 (AUC[0-24]) for MK-1496 Single Dose (21-Day Cycle)
Description: AUC[0-24] is a measure of the total plasma exposure of drug over a 24-hour period after the initial dose; for this analysis AUC was measured on Day 1 of the first 21-day cycle.
  AUC[0-24] for the 28-day cycle is reported as Outcome Measures 4 and 5.
Time Frame: Cycle 1, Day 1 (Hour 0 through Hour 24)
Population: All participants on the 21-day dosing schedule
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | MK-1496 20 mg (21-Day Cycle) | MK-1496 40 mg (21-Day Cycle) | MK-1496 80 mg (21-Day Cycle) | MK-1496 120 mg (21-Day Cycle)
Number analyzed (Participants) | 3 | 3 | 3 | 1
hr*nmol/L | 305 (246) | 434 (82.6) | 295 (193) | 1460

3. Secondary Outcome: Mean AUC[0-24] of MK-1496 on Day 1 of Multiple Dose Administration (28-Day Cycle)
Description: AUC is a measure of the total plasma exposure of a drug. For this analysis, AUC was measured just prior to dosing and through 24 hours postdose on Day 1 of Weeks 1, 2, and 3 in Cycle 1. The AUC value presented is the mean AUC for all measurements.
  AUC[0-24] for the Day 3 doses is reported as Outcome Measure 5.
Time Frame: Cycle 1, Day 1 (Hour 0 through Hour 24)
Population: All participants in the first cycle of the 28-day dosing schedule
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | MK-1496 20 mg (28-Day Cycle) | MK-1496 40 mg (28-Day Cycle) | MK-1496 80 mg (28-Day Cycle) | MK-1496 100 mg (28-Day Cycle) | MK-1496 120 mg (28-Day Cycle)
Number analyzed (Participants) | 3 | 3 | 6 | 2 | 3
hr*nmol/L | 122 (85.3) | 302 (47.7) | 936 (364) | 2530 (81.2) | 2320 (673)

4. Secondary Outcome: Mean AUC[0-24] of MK-1496 on Day 3 of Multiple Dose Administration (28-Day Cycle)
Description: AUC is a measure of the total plasma exposure of a drug. For this analysis, AUC was measured just prior to dosing and through 24 hours postdose on Day 3 of Weeks 1, 2, and 3 in Cycle 1. The AUC value presented is the mean AUC for all measurements.
  AUC[0-24] for the Day 1 doses is reported as Outcome Measure 4.
Time Frame: Cycle 1, Day 3 (Hour 0 through Hour 24)
Population: All participants in the first 28-day cycle
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Arm/Group | MK-1496 20 mg (28-Day Cycle) | MK-1496 40 mg (28-Day Cycle) | MK-1496 80 mg (28-Day Cycle) | MK-1496 100 mg (28-Day Cycle) | MK-1496 120 mg (28-Day Cycle)
Number analyzed (Participants) | 3 | 3 | 6 | 2 | 2
hr*nmol/L | 141 (114) | 366 (31.1) | 1300 (379) | 3090 (222) | 3470 (1560)

5. Primary Outcome: Number of Participants With Any Clinical or Laboratory Adverse Event
Description: This is a measure of the number of participants who experienced any adverse event (AE) while on study.
Time Frame: First dose up to 30 days after last dose (up to 2 years)
Population: All participants on study
Measure: Number; unit: participants
Arm/Group | MK-1496 20 mg (21-Day Cycle) | MK-1496 40 mg (21-Day Cycle) | MK-1496 80 mg (21-Day Cycle) | MK-1496 120 mg (21-Day Cycle) | MK-1496 20 mg (28-Day Cycle) | MK-1496 40 mg (28-Day Cycle) | MK-1496 80 mg (28-Day Cycle) | MK-1496 100 mg (28-Day Cycle) | MK-1496 120 mg (28-Day Cycle)
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 3 | 3 | 6 | 2 | 3
participants | 3 | 3 | 2 | 1 | 3 | 3 | 6 | 2 | 3

ADVERSE EVENTS:
Arm/Group | MK-1496 20 mg (21-Day Cycle) | MK-1496 40 mg (21-Day Cycle) | MK-1496 80 mg (21-Day Cycle) | MK-1496 120 mg (21-Day Cycle) | MK-1496 20 mg (28-Day Cycle) | MK-1496 40 mg (28-Day Cycle) | MK-1496 80 mg (28-Day Cycle) | MK-1496 100 mg (28-Day Cycle) | MK-1496 120 mg (28-Day Cycle)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/1 | 1/3 | 0/3 | 2/6 | 2/2 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 1/1 | 3/3 | 3/3 | 6/6 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1496 20 mg (21-Day Cycle) (N=3) | MK-1496 40 mg (21-Day Cycle) (N=3) | MK-1496 80 mg (21-Day Cycle) (N=3) | MK-1496 120 mg (21-Day Cycle) (N=1) | MK-1496 20 mg (28-Day Cycle) (N=3) | MK-1496 40 mg (28-Day Cycle) (N=3) | MK-1496 80 mg (28-Day Cycle) (N=6) | MK-1496 100 mg (28-Day Cycle) (N=2) | MK-1496 120 mg (28-Day Cycle) (N=3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1496 20 mg (21-Day Cycle) (N=3) | MK-1496 40 mg (21-Day Cycle) (N=3) | MK-1496 80 mg (21-Day Cycle) (N=3) | MK-1496 120 mg (21-Day Cycle) (N=1) | MK-1496 20 mg (28-Day Cycle) (N=3) | MK-1496 40 mg (28-Day Cycle) (N=3) | MK-1496 80 mg (28-Day Cycle) (N=6) | MK-1496 100 mg (28-Day Cycle) (N=2) | MK-1496 120 mg (28-Day Cycle) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 3 (3)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bactaermia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (3) | 1 (1)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts,or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.